CLINICAL TRIAL: NCT06334783
Title: Tumor Infiltrating Lymphocyte (TIL) Therapy for the Treatment of Advanced Solid Tumors
Brief Title: TIL for Patients With Advanced Solid Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio prioritization
Sponsor: Hervor Therapeutics (Industry)
Collaborators: Jinling Hospital, China (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HV-IIT
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TILs (Experimental): Biological: TILs Drug: IL-2
  Interventions: Biological: Autologous tumor-infiltrating lymphocyte cells

INTERVENTIONS:
Biological: Autologous tumor-infiltrating lymphocyte cells — On day 0, all patients will receive autologous tumor-infiltrating lymphocyte cells administered.

SUMMARY:
Background:

Tumor-infiltrating lymphocyte (TIL) therapy is a type of adoptive cellular therapy by harvesting infiltrated lymphocytes from tumors, culturing and amplifying them in vitro and then infusing back to patients.

TIL therapy has shown strong efficacy for the treatment of solid tumors and has achieved high objective response rates in multiple cancers, such as melanoma, NSCLC, and cervical cancer.

Objective:

To evaluate the safety and efficacy of TIL for the patients with advanced solid tumor.

Eligibility:

Adults aging 18-75 with advanced solid tumor.

Design:

1. Patients will undergo screening tests, including imaging procedures, heart and lung tests, and lab tests.
2. Freshly resected patient tumors were dissected by the surgeon.
3. TIL cells were isolated from the patient's tumor tissue, then cultured in vitro, activated and expanded.
4. At last TIL cells will be re-infused into the patients.

ELIGIBILITY:
Inclusion criteria:

1. Be able to understand and sign the Informed of Consent Document. Be willing to follow the procedure and protocol of the clinical trial.
2. Age ≥ 18 years and ≤ 75 years.
3. Expected survival time > 3 months.
4. ECOG score 0-1.
5. At least one lesion that could undergo surgery or biopsy to obtain tumor tissue for TIL preparation.
6. At least 1 measurable lesion (according to RECIST v1.1).
7. Metastatic or recurrent solid tumor, confirmed by histopathology. Patients who have failed previous standard treatment or currently do not have standard treatment, or who have been determined by the researcher to be unsuitable for current standard treatment due to other reasons.
8. Any previous anti-tumor treatment must exceed 28 days when collecting tumor tissue; The tumor tissue used for collecting and preparing TIL should not have undergone local treatment.
9. The bone marrow function of the subject's meets the following requirements:

   1. Absolute neutrophil count (ANC) ≥ 1.5× 10e9/L.
   2. Platelet (PLT） ≥ 75× 10e9/L.
   3. Hemoglobin (HGB) ≥ 90 g/L.
10. Liver and kidney function:

    1. Serum creatinine (Cr) ≤ 1.5 times of upper limit of normal (ULN) or creatine clearance ≥ 60 ml/min.
    2. Serum Alanine aminotransferase (ALT) or/and Aspartate aminotransferase (AST) ≤ 2.5 times of ULN.
    3. Total bilirubin (TBIL) ≤ 1.5 times of ULN.
11. Blood coagulation function:

    1. Prothrombin time (PT) ≤ 1.5 ULN.
    2. International Normalized Ratio (INR) ≤ 1.5 ULN.
    3. or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 ULN.
12. Left Ventricular Ejection Fractions (LVEF）≥45%.
13. Forced Expiratory Volume in the first second (FEV1）≥50%.
14. Women or men of childbearing potential should be ascetic or take contraception since the signing of ICF to 24 weeks or later after the last administration of drug.

Exclusion criteria:

1. Female subjects who are in pregnancy or lactation or have a positive baseline blood pregnancy test.
2. Individuals who have experienced severe allergic reactions to any drug or its components in this trial in the past.
3. Received any investigational medication within 28 days prior to TIL cell transfusion or participated in another clinical study at the same time.
4. History of other known malignant tumors within the previous 5 years.
5. Primary central nerve system (CNS) cancer, or Participants with CNS metastasis after localized treatment.
6. History or syndrome of autoimmune diseases.
7. History of immunodeficiency, including testing positive for Human Immunodeficiency Virus (HIV), or having other acquired or congenital immunodeficiency diseases.
8. Have a history of ≥ grade 3 thromboembolic events within the past 6 months or are currently receiving thrombolytic or anticoagulant treatment due to high risk of thrombosis.
9. History of hereditary or acquired hemorrhagic diseases.
10. Clinical cardiovascular diseases or symptoms.
11. Active infection present.
12. Active pulmonary tuberculosis infection.
13. positive hepatitis B surface antigen or positive hepatitis B core antibody or positive hepatitis C virus antibody.
14. Syphilis spirochete antibody positive.
15. Patients received major surgery or under severe injury within 28 days before TIL infusion.
16. Patients who received live vaccine or attenuated live vaccine 28 days before TIL infusion.
17. Patients who have drug addiction history, alcoholism, or drug users.
18. Patients who have previously received cell therapy (such as TCR-T, CAR-T, TIL, etc.)
19. Patients not suitable for the clinical trial evaluated by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Safety of TIL | Day 0 - Day 730
  The safety of TIL will be assessed based on the totality of dose-limiting toxicity (DLT) and adverse event (AE) data collected during this phase.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Day 0 - Day 730
  To evaluate the proportion of participants who have a confirmed partial response (PR) and complete response (CR) per RECIST v1.1 and iRECIST as assessed by the investigator.
Duration of Response (DOR) | Day 0 - Day 730
  To evaluate the duration from the time that criteria are met for CR or PR per RECIST v1.1 and iRECIST as assessed by the investigator until disease progression or death due to any cause.
Disease Control Rate (DCR) | Day 0 - Day 730
  To evaluate the percentage of participants with a best overall confirmed response of CR or PR at any time plus stable disease (SD) per RECIST v1.1 and iRECIST as assessed by the investigator.
Progression free survival (PFS) | Day 0 - Day 730
  To evaluate the time from the date of TIL infusion until disease progression per RECIST v1.1 and iRECIST as assessed by the investigator or death due to any cause.
Overall survival (OS) | Day 0 - Day 730
  To evaluate the time from the date of TIL infusion to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Nanjing Jinling Hospital, Nanjing, Jiangsu
  - Wowen's hospital, School of medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No